CLINICAL TRIAL: NCT06255496
Title: Evaluation of the Clinical Performance of the Quantra® System With the QStat® Cartridge in Obstetric Patients
Brief Title: QStat Cartridge in Obstetric Patients
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-048
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Blood Loss Massive; Post Partum Hemorrhage
Keywords: Quantra; Viscoelastic testing; Coagulation
MeSH Terms: conditions — Postpartum Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Obstetric Patients: Obstetric patient population at risk of experiencing excessive bleeding around the time of delivery
  Interventions: Diagnostic Test: Quantra Hemostasis Analyzer with the QStat Cartridge

INTERVENTIONS:
Diagnostic Test: Quantra Hemostasis Analyzer with the QStat Cartridge — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: Quantra System; QStat Cartridge

SUMMARY:
This study will assess the performance of the Quantra System with the QStat Cartridge versus standard of care coagulation testing in pregnant women at risk of bleeding at delivery.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The QStat Cartridge was developed to monitor hemostasis in patients that may experience a range of coagulopathies of various etiologies including fibrinolytic defects. These patients include the tobstetric hemorrhage population. The cartridge consists of four independent channels each containing different sets of reagents, which provide four measurements performed in parallel yielding five parameters that depict the functional status of a patient's coagulation system.

This multicenter, prospective, observational pilot study will evaluate the performance of the Quantra System with the QStat Cartridge as compared to standard of care coagulation testing in pregnant women at risk of bleeding at delivery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than18 years.
* Subject is pregnant or at least 24 h postpartum
* Conventional coagulation tests and/or viscoelastic testing are ordered for concern of possible coagulopathy based on one or more clinical scenarios including hemorrhage, suspected or confirmed placental abruption, amniotic fluid embolism, or placenta accreta spectrum
* Subject or subject's LAR is willing to provide informed consent, either prospectively or by deferred consent.

Exclusion Criteria:

* Subject is younger than 18 years old.
* Subject or subject's LAR is unwilling or unable to provide informed consent, either prospectively or by deferred consent.
* Subject is incarcerated at the time of the study.
* Subject is currently enrolled in a distinct study that might confound the results of the proposed study
* Subject is affected by a condition that, in the opinion of the clinical team, may pose additional risks

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females
Study Population: Parturients 18 years or older who are at risk of experiencing an obstetric hemorrhage around the time of delivery.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Comparison of Quantra Clot Time to laboratory aPTT test results | At the time hemorrhage is suspected, anticipated within 24 hours after birth
  Coagulation function assessed by Quantra Clot Time (CT, sec) and activated partial thromboplastin (aPTT, sec) test
Comparison of Quantra Fibrinogen Contribution to Clot Stiffness to laboratory coagulation fibrinogen test results | At the time hemorrhage is suspected, anticipated within 24 hours after birth
  Coagulation function assessed by Quantra Fibrinogen Contribution to Clot Stiffness (FCS, hPa) and Clauss fibrinogen (mg/dL) test
Comparison of Quantra Clot Time to ROTEM delta INTEM CT test results | At the time hemorrhage is suspected, anticipated within 24 hours after birth
  Coagulation function assessed by Quantra Clot Time (CT, sec) and ROTEM INTEM CT (sec) test
Comparison of Quantra Fibrinogen Contribution to Clot Stiffness to ROTEM delta FIBTEM test results | At the time hemorrhage is suspected, anticipated within 24 hours after birth
  Coagulation function assessed by Quantra Fibrinogen Contribution to Clot Stiffness (FCS, hPa) and ROTEM FIBTEM (mm) test

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Parkland Health, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No